CLINICAL TRIAL: NCT02763358
Title: Assessing the Bite Counter as a Tool for Food Intake Monitoring: Phase II
Brief Title: Assessing the Bite Counter
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00043670
Record Dates: First submitted 2016-04-08; First posted 2016-05-05 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-06

CONDITIONS: Weight Loss
Keywords: obesity; weight loss
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bites and Steps displayed (Other): All subjects will be assigned to one arm-daily bites and steps displayed on Bite Counter device
  Interventions: Device: Bite Counter

INTERVENTIONS:
Device: Bite Counter — This study is a 15-week assessment of the possible utility of a wrist-worn device, the Bite Counter, in assisting the weight loss behavior change efforts of overweight and obese individuals. The Bite Counter tracks and analyzes wrist motions to identify those associated with taking bites of food and drinking beverages. It also has a step-counter feature. This study is designed to determine if using the Bite Counter with specific goals to reduce the numbers of bites and increase the numbers of steps will result in those changes.

SUMMARY:
This study is designed to test the usability of the Bite Counter in an attempt to reduce participants' daily bites while also increasing their daily steps.

DETAILED DESCRIPTION:
Self-monitoring is an important component of behavioral management of obesity. The Bite Counter is a wrist-worn device which detects the motions characteristic of taking a bite of food or a drink of liquid, to provide the wearer with a cumulative count of bites and sips over the day. In earlier studies the method was shown to accurately count bites across a wide variety of foods, utensils and subject demographics, and to provide an unbiased intake measurement. The proposed work will continue to improve the bite counting method by adapting to varying eating rates, develop a self-managed bite count-based weight loss protocol, and perform an independent test of the protocol. An improved Bite Counter device will also measure activity (steps).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 18 and 70 (inclusive)
* Participants must have a BMI between 27 and 35
* Participants must have regular and reliable access to a Windows-based computer with an internet connection with USB connectivity
* Participants must be currently consuming at least 1400 calories per day
* Participants must demonstrate adequate compliance with using Bite Counter and uploading data during the two-week baseline period

Exclusion Criteria:

* Participants must have no history of any eating disorder
* Participants must not have participated in a weight loss program within the month prior to baseline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Reduction in the numbers of bites per day as displayed on the Bite Counter | 15 weeks

SECONDARY OUTCOMES:
Increase in the number of steps per day as displayed on the Bite Counter | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick O'Neil, PhD, Principal Investigator — Medical University of South Caolina
Locations (1):
- Medical University of South Carolina-Weight Management Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No